CLINICAL TRIAL: NCT00992498
Title: Effectiveness of Rehabilitation in COPD Outpatients With Comorbidities
Brief Title: Rehabilitation in Chronic Obstructive Pulmonary Disease Outpatients
Status: Completed | Type: Observational
Sponsor: Villa Pineta Hospital (Other)
Responsible Party: Principal Investigator, Prof. Clini Enrico, Professor, Villa Pineta Hospital
Other Study IDs: 02/2008
Record Dates: First submitted 2009-10-07; First posted 2009-10-09 (Estimated); Last update posted 2012-12-21 (Estimated); Status verified 2012-12

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD (Chronic Obstructive Pulmonary Disease); outpatients; rehabilitation; comorbidities; patient-centered outcome
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
A retrospective analysis on a cohort of unselected COPD patients admitted to pulmonary rehabilitation (PR) performed in one rehabilitation centre has shown that the usual program is feasible and effective even in the presence of complex comorbidities, although some combined diseases might reduce the overall proportion of patients who respond to pre-defined outcomes criteria (Crisafulli E, et al. Thorax 2008;63:487-92).

The aim of this prospective study is to describe the pattern of prevalence of the most frequently associated COPD-comorbidities and the clinical impact on rehabilitation outcomes, referred to 3 teaching and 1 private hospitals admitting for pulmonary rehabilitation purposes.

ELIGIBILITY:
Inclusion Criteria:

* Presence of COPD as defined and classified according to the Global Initiative for Chronic Obstructive Lung Disease (GOLD) guidelines
* Ability to perform a rehabilitation program.

Exclusion Criteria:

* Patients with asthma or any other pulmonary diseases (either obstructive or restrictive.
* Patients no able to complete a rehabilitation program

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: COPD outpatients eligible for pulmonary rehabilitation
Sampling Method: Non-Probability Sample
Enrollment: 316 (Actual)
Dates: Start 2008-01; Primary Completion 2008-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Nr. patients with a minimum clinically important difference (MCID) in quality of life (change in St George's Respiratory Questionnaire) | T0 (admission in hospital) - Tend (discharge, after 20 days)
Nr. patients with a minimum clinically important difference (MCID) in exercise tolerance (change in 6MWD) | T0 (admission in hospital) - Tend (discharge, after 20 days)
Nr. patients with a minimum clinically important difference (MCID) in breathless (change in MRC scale) | T0 (admission in hospital) - Tend (discharge, after 20 days)

SECONDARY OUTCOMES:
Percentage of patients who withdrew from rehabilitation. | Tend (discharge, after 20 days)
Prevalence of comorbidities associated to COPD | Tend (discharge, after 20 days)

CONTACTS AND LOCATIONS:
Overall Officials: Enrico M Clini, Prof., Principal Investigator — Villa Pineta Hospital and University of Modena
Locations (4):
- Italy (4):
  - Villa Pineta Hospital - University of Modena, Pavullo nel Frignano, Modena
  - Clinic Center Private Hospital, Naples
  - Dpt.of Clinical Sciences - University of Parma, Parma
  - Cardio-Thoracic Dpt - University of Pisa -, Pisa

REFERENCES:
- [Result] Crisafulli E, Costi S, Luppi F, Cirelli G, Cilione C, Coletti O, Fabbri LM, Clini EM. Role of comorbidities in a cohort of patients with COPD undergoing pulmonary rehabilitation. Thorax. 2008 Jun;63(6):487-92. doi: 10.1136/thx.2007.086371. Epub 2008 Jan 18. PMID 18203818
- [Derived] Crisafulli E, Gorgone P, Vagaggini B, Pagani M, Rossi G, Costa F, Guarriello V, Paggiaro P, Chetta A, de Blasio F, Olivieri D, Fabbri LM, Clini EM. Efficacy of standard rehabilitation in COPD outpatients with comorbidities. Eur Respir J. 2010 Nov;36(5):1042-8. doi: 10.1183/09031936.00203809. Epub 2010 Apr 22. PMID 20413540